CLINICAL TRIAL: NCT02775604
Title: Comparison of Home-based Video, Paper/Print Checklist and Professional Home Assessment in the Detection of Fall Hazards for Older Adults Living at Home: A Pilot Randomized Crossover Trial
Brief Title: Comparison of Home-based Video, Paper/Print Checklist and Professional Home Assessment in Detection of Fall Hazards at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HIREB 1950
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Identification of Home Fall Hazards
Keywords: fall risks at home; video technology; home assessment; distal radius fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Video (Other): GoPro Camera
  Interventions: Behavioral: Video based/Therapists' rating of comprehensive-home-fall-hazard-checklist (vt-CHFHC)
- Paper Checklist (Other): Homeowner Print Checklist
  Interventions: Behavioral: Paper based/Patient self-rating of comprehensive-home-fall-hazard-checklist (pp-CHFHC)

INTERVENTIONS:
Behavioral: Video based/Therapists' rating of comprehensive-home-fall-hazard-checklist (vt-CHFHC) — The participant will use GoPro technology and follow standardized instructions to inspect each room of their house. They will navigate through their home wearing the GoPro camera, recording images about their home and their usual activities and use a talk-aloud approach to describe what they are doing and seeing. The evaluator will provide no feedback during the assessments.
  Arms: Home-Based Video
Behavioral: Paper based/Patient self-rating of comprehensive-home-fall-hazard-checklist (pp-CHFHC) — A paper version of CHFHC and other self-reported documents will be completed by the participants in their homes based on standardized verbal instruction provided by the research staff.
  Arms: Paper Checklist

SUMMARY:
The purpose of this study is to assess the feasibility and potential impact of video analysis of footage taken with a GoPro camera video in comparison to a homeowner checklist or gold standard home assessment as a means of detecting home fall hazards.

Investigators hypothesize that the assessment of homes for fall hazards with a GoPro camera will be better than a homeowner paper checklist in hazard identification.

DETAILED DESCRIPTION:
80 community-dwelling adults (50-75 years of age) will be recruited from clinics and the community through posters and advertising (n = 40 in the Healthy Group; n = 40 in the Distal Radius Fracture (DRF) Group (adults with 3-12 months post-DRF)).

Participants will be randomly allocated to a homeowner paper checklist or a GoPro video assessment and then cross-over to the opposite intervention.

To assess accuracy, a gold standard home assessment will be completed by a trained evaluator, after the homeowner checklist and GoPro video assessment.

Upon completion of the data collection, the evaluator will conduct their assessment (gold standard); review the findings from the GoPro "playback" with the participant, and conduct a semi-structured interview on their prior awareness of fall hazards, perceptions about the different methods of detecting fall hazards in their home; and intentions to remediate identified hazards.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Group: community-dwelling adults
* DRF Group: adults with 3-12 months post DRF
* ability to read, understand and speak English

Exclusion Criteria:

* identified cognitive disorder
* major loss of vision or hearing
* other concurrent upper extremity injuries or neurological impairments
* any unhealed fractures

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation Agreement | Within 1 week of completion of assessment
  Fall hazard scores will be calculated based on the number and severity of hazards identified from the paper checklist, the GoPro assessment, and the independent evaluation. The extent of agreement on fall-hazard score and time taken to complete the evaluations (home-based video, paper/print checklist; professional home assessment) will be assessed.

SECONDARY OUTCOMES:
Feasibility and Fidelity | Within 1 week of completion of assessment
  Semi-structured phone interviews will be conducted to collect participant feedback on the feasibility, usability, usefulness, acceptance, barriers, facilitators, respondent burden and preference for using GoPro video-technology vs. pp-CHFHC vs. professional assessment. During the interview, participants will also be asked about their prior awareness of fall hazards and experiences about the different methods of detecting fall hazards in their home.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No